CLINICAL TRIAL: NCT01017068
Title: Aqueous Mushroom Extract as a Glaucoma Agent
Brief Title: Aqueous Mushroom Extract and Intraocular Pressure
Acronym: AME
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Benin (Other)
Responsible Party: Prof. V.I, Iyawe, Dean, College of Basic Medical Sciences. UNIBEN.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRLLSAW
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Glaucoma
Keywords: GLAUCOMA
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A1 (glaucoma) (Experimental)
  Interventions: Drug: OME
- A2 (glaucoma) (Experimental)
  Interventions: Drug: OME
- A3 (glaucoma) (Experimental)
  Interventions: Drug: OME
- A1 (normals) (Experimental)
  Interventions: Drug: OME
- A2 (normals) (Experimental)
  Interventions: Drug: OME
- A3 (normals) (Experimental)
  Interventions: Drug: OME

INTERVENTIONS:
Drug: OME — 4g/100ml) dose: п gutt tid x 1/52
  Arms: A1 (glaucoma)
Drug: OME — (2g/100ml) dose: п gutt tid x 1/52
  Arms: A2 (glaucoma)
Drug: OME — (1g/100ml) dose: п gutt tid x 1/52
  Arms: A3 (glaucoma)
Drug: OME — (4g/100ml) dose: п gutt tid x 1/52
  Arms: A1 (normals)
Drug: OME — (2g/100ml) dose: п gutt tid x 1/52
  Arms: A2 (normals)
Drug: OME — (1g/100ml) dose: п gutt tid x 1/52
  Arms: A3 (normals)

SUMMARY:
The purpose of this study is to determine the effect of Aqueous mushroom extract (AME) on intra ocular pressure (IOP) in humans or as a potential anti glaucoma drug.

DETAILED DESCRIPTION:
The Prophet of Islam (Peace Be On Him) was reported to have said that 'mushroom are like manna and their water heals eye diseases'(Sahih Bukhari 1985). This statement is being investigated in view of the link between blood pressure and intra ocular pressure.

Glaucoma which is a sight threatening disease and is associated with raised intraocular pressure has been treated for a long time with beta blockers. Nowadays the drugs of choice are prostaglandin analogs. This study seeks to discover the effect of pleurotus tuberregium on raised intraocular pressure and to compare its effect on I.O.P with that of known glaucoma drugs. This study also seeks to find out at what concentration pleurotus is effective significantly on raised intraocular pressure

Clinical Investigation will be conducted in the Ophthalmological unit of UBTH in two phases. In the first phase 21 relatively young healthy subjects aged less than 50 yrs will be recruited for this study after their informed consent. They will have no previous systemic or ocular diseases and have an intraocular pressure of 19mmHg or less and a visual acuity of 6/6. Base line investigations will include the systolic and diastolic blood pressure, horizontal pupillary diameter and applanation tonometry. The subjects will be divided into three groups of seven each (A1, A2 and A3).

The study will at first constitute two weeks mushroom treatment, two weeks no mushroom treatment and then two weeks mushroom treatment. Treatment will be with aqueous extract of Oyster Medicinal mushroom Extract (4g/100ml) dose: п gutt tid x 1/52 for A1, 2g/100ml dose: п gutt tid x 1/52 for A2 and 1g/100ml dose: п gutt tid x 1/52 for A3. Investigations of the baseline parameters will be done at the start and after each seven days. The subjects will be monitored to ensure full compliance with the designed protocol.

The second phase will involve an equal number of age matched ocular hypertensive or glaucoma patient undergoing treatment in UBTH. They will also be divided into three groups of seven each and the treatment regimen above repeated. The IOP in this case will be taken by a masked observer.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of open angle glaucoma
* intraocular pressure above 23mmHg

Exclusion Criteria:

* close angle glaucoma
* end stage of glaucoma visual field loss
* ocular disease other than glaucoma that will interfere with result

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-02 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
DECREASE INTRA OCULAR PRESSURE | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: VINCENT I IYAWE, MD, PhD, Study Chair — University of Benin, Benin City Nigeria
Locations (1):
- Eye Clinic University of Benin Teaching Hospital, Benin City, Edo, Nigeria

REFERENCES:
- [Background] Akinlabi GA, Igbinigie EV, Akpaja EO, Iyawe VI. Preliminary study on the effect of medicinal mushroom extract and timolol maleate on dexamethasone induced ocular hypertension in feline's eye model.Journal of Medicine and Biomedical Research 6(2)63-68. Akinlabi GA, Uzibor HI, Iyawe IO, Iyawe VI. Effect of oyster mushroom exract(pleurotus ostreatus) and latanoprost on intra ocular pressure using cat's eye model. Journal of Medicine and Biomedical Research 8(1)58-64.